CLINICAL TRIAL: NCT04851171
Title: A Randomized Controlled Trial Comparing Semi-rigid Ureteroscopy and Flexible Ureteroscopy For the Treatment of Proximal Ureteric Stone
Brief Title: Semi-rigid Ureteroscopy Versus Flexible Ureteroscopy For the Treatment of Proximal Ureteric Stone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Ibrahim Alnadhari, Associate Consultant- Surgery, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-19-036
Record Dates: First submitted 2021-04-01; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Ureteric Stone; Stone Ureter
Keywords: Urolithiasis; Ureteroscopy; Ureteric stone; Flexible ureteroscopy; Semi-rigid ureteroscopy
MeSH Terms: conditions — Ureterolithiasis; Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-rigid Ureteroscopy (Active Comparator): Patient with upper ureteric stone who are randomized in this arm will undergo semi-rigid ureteroscopy for treatment of the stone.
  Interventions: Procedure: Semi-rigid Ureteroscopy
- Flexible Ureteroscopy (Active Comparator): Patient with upper ureteric stone who are randomized in this arm will undergo flexible ureteroscopy for treatment of the stone.
  Interventions: Procedure: Flexible Ureteroscopy

INTERVENTIONS:
Procedure: Flexible Ureteroscopy — Flexible ureteroscopy is the use of flexible ureteroscope for the treatment of stone in the upper ureter with the aid of laser lithotripsy.
  Arms: Flexible Ureteroscopy
Procedure: Semi-rigid Ureteroscopy — Semi-rigid ureteroscopy is the use of the semi-rigid ureteroscope for the treatment of stone in the upper ureter with the aid of laser lithotripsy.
  Arms: Semi-rigid Ureteroscopy

SUMMARY:
The present study is randomized in nature, comparing the stone free rate and complications rate between semi-rigid ureteroscopy (SR-URS) and Flexible Ureteroscopy (F-URS) for the treatment of Proximal Ureteric stone (PUS), whereby the preoperative assessments, procedure and reporting of outcomes will all be standardized.

DETAILED DESCRIPTION:
There are various treatment options that can be used for the treatment of PUS, which include extracorporeal shockwave lithotripsy (SWL), ureteroscopy (URS), percutaneous nephrolithotomy (PCNL), antegrade uretero-lithotripsy, laparoscopy, and rarely, open surgical procedures. However, the standard, and the most frequently used modalities are SWL and ureteroscopy. When comparing the effectiveness in the treatment of Proximal Ureteric stone (PUS) between SWL and URS, SWL has lower rates of complication and morbidity, but URS has a higher likelihood of successfully treating the patient within a single procedure. Additionally, with the advancements in technology and miniaturization of the ureteroscopes, along with the presence of auxiliary instruments such as holmium laser and retrieval baskets, ureteroscopy is more widely used.

In the proximal ureter, SR-URS tends to encounter difficulties in accessing the stone, but F-URS aids in overcoming those difficulties. As a result, the use of F-URS for PUS has indicated a strong success rate with lower likelihood of complications. When comparing the drawbacks of the two types of modalities, F-URS tends to be more expensive, and requires auxiliary instruments. And SR-URS tends to have lower success rate along with an increased rate in complications.

The precedence of FURS over SR-URS in the treatment of PUS is yet to be extensively studied. Presently there are only five studies that have compared the two modalities of treatment. But, due to the lack standardization of variables, procedure, follow-up imaging and reporting of outcomes in the past studies, it is imperative to conduct study that is prospective and randomized in nature.

The present study is randomized in nature, comparing the stone free rate and complications rate between SR-URS and F-URS for the treatment of PUS, whereby the preoperative assessments, procedure and reporting of outcomes will all be standardized.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Single proximal ureteric stone indicated for active treatment with ureteroscopy (stented or non-stented)

Exclusion Criteria:

* Solitary Kidney
* Bilateral ureteric stones
* Ipsilateral multiple simultaneous ureteric stones
* Ipsilateral kidney stone
* Active UTI
* Coagulopathy diseases
* Ipsilateral ureteral anomalies, ureteral disorder (tumor or stricture) or previous ureteral open surgery.
* Pregnant patients.
* Unable to give informed consent.
* Patient is not agreeing to go through the randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | Four weeks
  Sone free status will be assessed by doing CT KUB scan 4 weeks postoperative and it is defined as patients with no residual stones or clinically insignificant residual fragments (< 2 mm).

SECONDARY OUTCOMES:
Complication rate | Three Months
  To evaluate the complication rate post procedure including infection rate, genitourinary injury, hematuria, emergency visits rate and we will use of modified Calvin Dindo classification to grade the surgical complications.
To compare stone free rate and complications between patients with ureteric stent and patients without ureteric stent | Three Months
  Patients will be stratified into two groups: group 1 with ureteric stents and group 2 without ureteric stents. Then comparison between the two groups in regards the stone free rate and the complications rate as per the previous definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Al-Nadhari, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Al Wakra Hospital, Al-Wakrah, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf JS Jr. Treatment selection and outcomes: ureteral calculi. Urol Clin North Am. 2007 Aug;34(3):421-30. doi: 10.1016/j.ucl.2007.04.010. PMID 17678991
- [Background] Lee JH, Woo SH, Kim ET, Kim DK, Park J. Comparison of Patient Satisfaction with Treatment Outcomes between Ureteroscopy and Shock Wave Lithotripsy for Proximal Ureteral Stones. Korean J Urol. 2010 Nov;51(11):788-93. doi: 10.4111/kju.2010.51.11.788. Epub 2010 Nov 17. PMID 21165201
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART II. J Urol. 2016 Oct;196(4):1161-9. doi: 10.1016/j.juro.2016.05.091. Epub 2016 May 27. PMID 27238615
- [Background] Hyams ES, Monga M, Pearle MS, Antonelli JA, Semins MJ, Assimos DG, Lingeman JE, Pais VM Jr, Preminger GM, Lipkin ME, Eisner BH, Shah O, Sur RL, Mufarrij PW, Matlaga BR. A prospective, multi-institutional study of flexible ureteroscopy for proximal ureteral stones smaller than 2 cm. J Urol. 2015 Jan;193(1):165-9. doi: 10.1016/j.juro.2014.07.002. Epub 2014 Jul 9. PMID 25014576
- [Background] Alkan E, Saribacak A, Ozkanli AO, Basar MM, Acar O, Balbay MD. Flexible Ureteroscopy Can Be More Efficacious in the Treatment of Proximal Ureteral Stones in Select Patients. Adv Urol. 2015;2015:416031. doi: 10.1155/2015/416031. Epub 2015 Nov 4. PMID 26617636
- [Background] Galal EM, Anwar AZ, El-Bab TK, Abdelhamid AM. Retrospective comparative study of rigid and flexible ureteroscopy for treatment of proximal ureteral stones. Int Braz J Urol. 2016 Sep-Oct;42(5):967-972. doi: 10.1590/S1677-5538.IBJU.2015.0644. PMID 27622276
- [Background] Karadag MA, Demir A, Cecen K, Bagcioglu M, Kocaaslan R, Altunrende F. Flexible ureterorenoscopy versus semirigid ureteroscopy for the treatment of proximal ureteral stones: a retrospective comparative analysis of 124 patients. Urol J. 2014 Nov 1;11(5):1867-72. PMID 25361706